CLINICAL TRIAL: NCT00482170
Title: A 3 Month, Randomised, Open Label, Parallel Group, Descriptive Study to Explore and Compare Perceptions and Satisfaction for Two Different Delivery Mechanisms for Etanercept (Etanercept Auto-injector and the Etanercept Prefilled Syringe) in Patients With Psoriasis.
Brief Title: Compare Perceptions and Satisfaction for Two Different Delivery Mechanisms for Etanercept
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881A6-3326
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

ARMS (2):
- 1 (Experimental): Arm 1: Enbrel 50 mg Prefilled Syringe
  Interventions: Device: Enbrel (etanercept)
- 2 (Active Comparator): Arm 2 Enbrel 50 mg Autoinjector
  Interventions: Device: Etanercept

INTERVENTIONS:
Device: Enbrel (etanercept) — Arm 1 = Enbrel 50 mg Prefilled Syringe twice weekly
  Arms: 1
Device: Etanercept — Arm 2 = Enbrel 50 mg Autoinjector twice weekly
  Arms: 2

SUMMARY:
Primary objective of this study is to compare patient satisfaction with the prefilled syringe (PFS) and the auto-injector (AI), two different delivery devices for etanercept after 12 weeks of use, using a 10 point scale form totally dissatisfied to totally satisfied.Secondary evaluation focus on the identification of patient and device attributes associated with patient satisfaction.

DETAILED DESCRIPTION:
For the measures of patient's satisfaction with and perceptions of, their device, standard Likert scales are used. This allows the magnitude of individual's perceptions and satisfaction to be measured on a multipoint scale anchored at each end. In addition, the study will describe patient perceptions related to device attributes, which are of importance in describing overall patient perception. A range of potential device benefits (e.g. ease of use, convenience, injection site pain, injection anxiety, injection confidence) will be captured using a questionnaire. The study aims to characterize patient attributes that will indicate when one device may result in greater patient satisfaction than another. Patient attributes are composed of patient characteristics (e.g. age, sex, demographics, social and educational status psychological status, willingness to self-manage, injection experience) and Psoriasis characteristics (e.g. disease severity, disease duration, co morbidities, prior treatment, quality of life). The study will also take the opportunity to measure health outcome measures as there may be important differences in cost of training and patient support between the two devices.

ELIGIBILITY:
Inclusion Criteria:

* Treatment of adults with moderate to severe plaque psoriasis who failed to respond to, or who have a contraindication to, or are intolerant to other systemic therapy including cyclosporine, methotrexate or PUVA
* Eligible for treatment with etanercept according to Summary of Product Characteristics (SmPC), and applicable local guidelines.
* Aged 18 years or more
* Willing and able to self-inject etanercept.
* Able to store test drug at 2-8oC.
* Negative serum ß-human chorionic gonadotropin (ß-HCG) pregnancy test at baseline (week 0) for all women of childbearing potential. Sexually active women of childbearing potential must use a medically acceptable form of contraception. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices, or properly used barrier contraception. Sexually active men must agree to use a reliable form of contraception during the study.
* Capable of understanding and willing to provide signed and dated written voluntary informed consent before any protocol-specific procedures are performed.

Exclusion Criteria:

* Prior experience of biologics and anti-TNF treatment for their Psoriasis including etanercept.
* Sepsis or risk of sepsis.
* Current or recent infections, including chronic or localized.
* Latex sensitivity.
* Vaccination with live vaccine in last 4 weeks, or expected to require such vaccination during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (72):
- Belgium (7):
  - Bruges
  - Brussels
  - Edegem
  - Ghent
  - Hasselt
  - Kapellen
  - Liège
- Denmark (3):
  - Hellerup
  - Hørsholm
  - Roskilde
- Finland (3):
  - Helsinki
  - Joensuu
  - Tampere
- France (10):
  - Le Mans, Cedex
  - Limoges
  - Montpellier
  - Nancy
  - Nantes
  - Paris
  - Pessac
  - Pierre-Bénite
  - Reims
  - Toulouse
- Germany (19):
  - Augsburg
  - Berlin
  - Bonn
  - Cologne
  - Dresden
  - Dülmen
  - Erlangen
  - Freiburg im Breisgau
  - Göttingen
  - Greifswald
  - Hamburg
  - Lübeck
  - Mainz
  - Mannheim
  - München
  - Münster
  - Tübingen
  - Wiesbaden
  - Würzburg
- Greece (3):
  - Athens
  - Ioannina
  - Thessaloniki
- Szeged, Hungary
- Italy (10):
  - S. Giovanni Rotondo, Foggia
  - Terracina, Latina
  - Gallarate, Varese
  - Capranica, Viterbo
  - Bologna
  - Como
  - Milan
  - Napoli
  - Padua
  - Pisa
- Netherlands (3):
  - Breda
  - Flushing
  - Nijmegen
- Norway (3):
  - Bergen
  - Stavanger
  - Tromsø
- Spain (6):
  - Elche, Alicante
  - Santander, Cantabria
  - Córdoba
  - Granada
  - Madrid
  - Valencia
- Sweden (4):
  - Danderyd
  - Gothenburg
  - Linköping
  - Malmo

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept 50 mg Auto-injector: Etanercept (Enbrel) 50 milligram (mg) auto-injector (AI) subcutaneously (s.c.) twice-weekly for 12 weeks.
- Etanercept 50 mg Prefilled Syringe: Etanercept (Enbrel) 50 mg prefilled syringe (PFS) s.c. twice-weekly for 12 weeks.
Period: Overall Study
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Started | 207 | 214
Treated | 207 | 211
Completed | 192 | 194
Not Completed | 15 | 20
Not completed — Adverse Event | 5 | 14
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Protocol Violation | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Unspecified reason | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Etanercept 50 mg Auto-injector: Etanercept (Enbrel) 50 mg AI s.c. twice-weekly for 12 weeks.
- Etanercept 50 mg Prefilled Syringe: Etanercept (Enbrel) 50 mg PFS s.c. twice-weekly for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe | Total
Number analyzed (Participants) | 206 | 211 | 417
Age Continuous [Mean (Standard Deviation); unit: years] — Out of a total of 421 participants, data for baseline measure (age) was available for 417 participants who were treated and had at least 1 efficacy evaluation.
  years | 46.1 (13.2) | 46.1 (13.4) | 46.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Out of a total of 421 participants, data for baseline measure (gender) was available for 417 participants who were treated and had at least 1 efficacy evaluation.
  Participants
    Female | 71 | 65 | 136
    Male | 135 | 146 | 281

OUTCOME MEASURES:

1. Primary Outcome: Participant Satisfaction With Injection Device Evaluated at Week 12 for Modified Intent-to-treat (mITT) Population
Description: Participant satisfaction was assessed by asking the question, "How satisfied are you with your injection device?" using a 0-10 point scale, where 0= totally dissatisfied and 10= totally satisfied.
Time Frame: Week 12
Population: Modified intent-to-treat (mITT) analysis population included all randomized participants who received at least 1 injection of study medication and had at least 1 efficacy evaluation. Here, 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 198 | 197
units on a scale | 8.9 (1.9) | 7.6 (2.6)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Analysis of variance (ANOVA) using mixed linear model with participant as random effect, treatment group, visit and the interaction between treatment group and visit as fixed factors and with an unstructured correlation was used for the analysis; Test type: Non-Inferiority or Equivalence — The non-inferiority test was performed using the 95 percent (%) confidence interval (CI) of the difference of mean participant satisfaction (alpha = 2.5%). Non-inferiority was demonstrated if the lower limit of the 2-sided CI is greater than -1; p < 0.001, ANOVA — Statistical testing, one-sided, was done at 2.5% significance level; Mean Difference (Final Values) = 1.32, 95% CI 2-sided [0.87 to 1.77], Standard Error of Mean 0.23

2. Primary Outcome: Participant Satisfaction With Injection Device at Week 12 for Per-protocol (PP) Population
Description: as for outcome 1
Time Frame: Week 12
Population: Per-protocol (PP) analysis population included participants from mITT population who completed the study with no major protocol violations. Here, 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 189 | 186
units on a scale | 9.0 (1.9) | 7.5 (2.6)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; ANOVA using a mixed linear model with participant as random effect, treatment group, visit and the interaction between treatment group and visit as fixed factors and with an unstructured correlation was used for the analysis; Test type: Non-Inferiority or Equivalence — The non-inferiority test was performed using the 95% CI of the difference of mean participant satisfaction (alpha = 2.5%). Non-inferiority was demonstrated if the lower limit of the 2-sided CI is greater than -1; p < 0.001, ANOVA — Statistical testing, one-sided, was done at 2.5% significance level; Mean Difference (Final Values) = 1.41, 95% CI 2-sided [0.95 to 1.87], Standard Error of Mean 0.23

3. Secondary Outcome: Percentage of Participants Satisfied With Injection Device
Description: Participant satisfaction was assessed by asking the question "Are you satisfied with your injection device? and using a dichotomous response: Yes or No.
Time Frame: Baseline, Week 4 and Week 12
Population: mITT analysis population included all randomized participants who received at least 1 injection of study medication and had at least 1 efficacy evaluation. 'n' is signifying those participants who were evaluated for this measure at the time point for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
percentage of participants
  Baseline- After the training (n=198, 199) | 99.5 | 92.5
  Week 4 (n=190, 190) | 98.9 | 90.0
  Week 12 (n=188, 179) | 98.4 | 88.8
  Last Observation (n=206, 210) | 98.5 | 88.6
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Baseline- after the training: Generalized Estimating Equations (GEE) model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment group, visit and the interaction between treatment group and visit as fixed factors was used for the analysis; Test type: Superiority or Other; p = 0.008, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 16.12, 95% CI 2-sided [2.05 to 126.9]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Week 4: GEE model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment group, visit and the interaction between treatment group and visit as fixed factors was used for the analysis; Test type: Superiority or Other; p = 0.002, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 11.25, 95% CI 2-sided [2.44 to 51.83]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Week 12: GEE model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment group, visit and the interaction between treatment group and visit as fixed factors was used for the analysis; Test type: Superiority or Other; p = 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 7.88, 95% CI 2-sided [2.26 to 27.44]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Last observation: Logistic regression was used for the analysis; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 8.73, 95% CI 2-sided [2.59 to 29.47]

4. Secondary Outcome: Influence of Age on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the delivery mechanism. Age categories were defined based on quartiles (Q) of ages observed. Participants were divided into quarters: less than or equal to (=<) 36 years, greater than (>) 36 years to 45 years, > 45 years to 55 years, > 55 years.
Time Frame: Week 12
Population: mITT analysis population included all randomized participants who received at least 1 injection of study medication and had at least 1 efficacy evaluation. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  =< 36 years | 8.94 (1.95) | 7.18 (2.62)
  > 36 years to 45 years | 8.91 (1.52) | 7.41 (2.39)
  > 45 years to 55 years | 9.06 (1.89) | 7.93 (2.90)
  > 55 years | 8.82 (2.12) | 8.07 (2.49)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between all categories, by 10 unit increment. Univariate model in which all continuous variables were considered continuous and mean centered was used; Test type: Superiority or Other; p = 0.045, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = 0.17, 95% CI 2-sided [0.00 to 0.34]

5. Secondary Outcome: Influence of Gender on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the delivery mechanism. Gender categories were defined as male and female.
Time Frame: Week 12
Population: mITT analysis population included all randomized participants who received at least 1 injection of study medication and had at least 1 efficacy evaluation. LOCF method was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Male | 9.07 (1.59) | 7.60 (2.57)
  Female | 8.70 (2.31) | 7.68 (2.66)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between categories, female and male (reference); Test type: Superiority or Other; p = 0.707, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = -0.09, 95% CI 2-sided [-0.58 to 0.39]

6. Secondary Outcome: Influence of Socio-educational Status on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the delivery mechanism. Socio-educational status categories were defined as reading or (/) writing capacity, high school /baccalaureate level and university level.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Reading /Writing capacity | 9.22 (1.62) | 7.96 (2.49)
  High school /Baccalaureate level | 8.80 (1.97) | 7.55 (2.73)
  University level | 8.89 (2.01) | 7.24 (2.39)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between categories, high school or baccalaureate level and reading or writing capacity (reference); Test type: Superiority or Other; p = 0.195, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = -0.38, 95% CI 2-sided [-0.89 to 0.14]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between categories, university level and reading or writing capacity (reference); Test type: Superiority or Other; p = 0.195, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = -0.55, 95% CI 2-sided [-1.21 to 0.11]

7. Secondary Outcome: Influence of Psychological Status as Assessed by Hospital Anxiety Depression (HAD) Score on Participant Satisfaction With Injection Device
Description: Participant satisfaction scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher score = greater satisfaction with injection device. Psychological status was assessed using participant rated questionnaire with 2 subscales for anxiety (HAD-A) and depression (HAD-D). Total score: 0 to 21 for each subscale; higher score = greater severity of symptoms. Score categories were based on quartiles of HAD-A and HAD-D scores observed. Participants were divided into quarters: =< 4, > 4 to 7, > 7 to 10, > 10 for HAD-A and =< 3, > 3 to 5, > 5 to 8, > 8 for HAD-D.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  HAD-A: =< 4 | 8.98 (1.77) | 7.83 (2.42)
  HAD-A: > 4 to 7 | 9.17 (1.48) | 7.49 (2.65)
  HAD-A: > 7 to 10 | 8.89 (2.27) | 7.42 (2.88)
  HAD-A: > 10 | 8.73 (1.92) | 7.74 (2.44)
  HAD-D: =< 3 | 8.68 (2.19) | 7.93 (2.39)
  HAD-D: > 3 to 5 | 9.15 (2.04) | 7.57 (2.42)
  HAD-D: > 5 to 8 | 9.20 (1.02) | 7.50 (2.50)
  HAD-D: > 8 | 8.90 (1.92) | 7.31 (3.09)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between categories, HAD-A: =< 4, HAD-A: > 4 to 7, HAD-A: > 7 to 10 and HAD-A: > 10; by 5 unit increment. Univariate model in which all continuous variables were considered continuous and mean centered was used; Test type: Superiority or Other; p = 0.493, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = -0.09, 95% CI 2-sided [-0.36 to 0.17]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between categories, HAD-D: =< 3, HAD-D: > 3 to 5, HAD-D: > 5 to 8 and HAD-A: > 8; by 5 unit increment. Univariate model in which all continuous variables were considered continuous and mean centered was used; Test type: Superiority or Other; p = 0.287, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = -0.16, 95% CI 2-sided [-0.46 to 0.14]

8. Secondary Outcome: Influence of Willingness to Self Manage as Assessed by Patient Activation Measure (PAM) on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the injection device. The 13-item short form of the PAM survey assessed participants' knowledge, skill, and confidence for self-management; calibrated scale score ranged from 0 to 100. Higher scores indicated more confidence in managing participants' condition and lifestyle. Score categories were defined based on quartiles of PAM scores observed. Participants were divided into quarters: =< 47.4, > 47.4 to 56.4, > 56.4 to 68.5, > 68.5.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  =< 47.4 | 8.73 (1.90) | 7.05 (2.76)
  > 47.4 to 56.4 | 9.41 (1.14) | 7.94 (2.17)
  > 56.4 to 68.5 | 8.28 (2.68) | 7.94 (2.70)
  > 68.5 | 9.11 (1.73) | 7.93 (2.49)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.123, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = 0.13, 95% CI 2-sided [-0.04 to 0.30]

9. Secondary Outcome: Influence of Prior Self-injection Experience on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the injection device. The categories were defined based on presence of any prior experience of self-injection. Participants were divided into categories: yes and no.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Yes | 8.89 (1.92) | 7.53 (2.74)
  No | 8.96 (1.87) | 7.66 (2.53)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between categories, yes and no (reference); Test type: Superiority or Other; p = 0.359, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = -0.24, 95% CI 2-sided [-0.76 to 0.28]

10. Secondary Outcome: Influence of Duration of Psoriasis on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the injection device. Duration of psoriasis categories were defined based on quartiles of the duration of psoriasis observed. Participants were divided into quarters: =< 11 years, > 11 years to 19 years, > 19 years to 28 years, > 28 years.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  =< 11 years | 9.09 (1.56) | 7.90 (2.22)
  > 11 years to 19 years | 8.74 (1.99) | 7.17 (2.67)
  > 19 years to 28 years | 9.12 (1.65) | 7.72 (2.76)
  > 28 years | 8.82 (2.29) | 7.76 (2.66)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between all categories, by 5 unit increment. Univariate model in which all continuous variables were considered continuous and mean centered was used; Test type: Superiority or Other; p = 0.693, Regression, Linear; Regression coefficient = 0.02, 95% CI 2-sided [-0.08 to 0.12]

11. Secondary Outcome: Influence of Physician Global Assessment (PGA) of Psoriasis on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the injection device. PGA of Psoriasis scale ranges from 0 (no psoriasis) to 5 (severe disease). 'Clear' and 'Almost clear' includes all participants who were scored as a 0 or 1. Score categories were defined based on quartiles of PGA scores observed. Participants were divided into: =< 3, > 3 to 4, > 4.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  =< 3 | 8.87 (1.91) | 7.51 (2.48)
  > 3 to 4 | 8.96 (1.97) | 7.79 (2.79)
  > 4 | 9.62 (0.51) | 7.83 (3.06)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between all categories, by 1 unit increment. Univariate model in which all continuous variables were considered continuous and mean centered was used; Test type: Superiority or Other; p = 0.170, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = 0.22, 95% CI 2-sided [-0.09 to 0.53]

12. Secondary Outcome: Influence of Psoriasis Area and Severity Index (PASI) on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the injection device. PASI: combined assessment of lesion severity and area affected into single score; range: 0= no disease to 72= maximal disease. Score categories were defined based on quartiles of PASI score observed. Participants were divided into quartiles: =< 11.2, > 11.2 to 16.2, > 16.2 to 21.9, > 21.9.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  =< 11.2 | 8.41 (2.26) | 7.45 (2.33)
  > 11.2 to 16.2 | 9.17 (1.97) | 7.81 (2.78)
  > 16.2 to 21.9 | 9.11 (1.66) | 7.67 (2.49)
  > 21.9 | 9.00 (1.57) | 7.67 (2.79)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.211, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = 0.02, 95% CI 2-sided [-0.01 to 0.04]

13. Secondary Outcome: Influence of Participant's Assessment of General Health on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the injection device. Participant's assessment of general health was measured on 100 millimeter (mm) line visual analog scale (VAS). 0 mm = extremely bad to 100 mm = very well. Score categories were defined based on quartiles of VAS score observed. Participants were divided into quarters: =< 48, > 48 to 67.25, > 67.25 to 84, > 84.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  =< 48 | 8.54 (2.36) | 7.06 (3.26)
  > 48 to 67.25 | 9.15 (1.24) | 7.79 (2.61)
  > 67.25 to 84 | 8.70 (2.22) | 7.72 (2.06)
  > 84 | 9.42 (1.20) | 7.85 (2.44)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.045, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = 0.09, 95% CI 2-sided [0.00 to 0.18]

14. Secondary Outcome: Influence of Participant's Global Assessment of Psoriasis on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the injection device. Participant's global assessment of psoriasis was measured using a 100 mm VAS, with 0 = no activity and 100 = extremely active psoriasis. Score categories were defined based on quartiles of participant's global assessment of psoriasis scores observed. Participants were divided into quarters: =< 63, > 63 to 76, > 76 to 88, > 88.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  =< 63 | 8.79 (1.54) | 7.96 (2.18)
  > 63 to 76 | 9.02 (1.91) | 7.51 (2.80)
  > 76 to 88 | 8.71 (2.19) | 7.70 (2.55)
  > 88 | 9.20 (1.90) | 7.33 (2.78)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.913, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = -0.01, 95% CI 2-sided [-0.12 to 0.11]

15. Secondary Outcome: Influence of Dermatology Life Quality Index (DLQI) on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the injection device. DLQI is the dermatology-specific quality of life measure used for psoriatic population. The 10-item questionnaire has a score range of 0 to 30 with higher scores indicating poor quality of life. Score categories were defined based on quartiles of DLQI scores observed. Participants were divided into quarters: =< 8, > 8 to 13, > 13 to 18, > 18.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  =< 8 | 8.82 (2.18) | 7.82 (2.23)
  > 8 to 13 | 8.94 (1.70) | 7.71 (2.53)
  > 13 to 18 | 8.81 (2.04) | 7.37 (2.72)
  > 18 | 9.14 (1.67) | 7.55 (2.87)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.968, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = -0.00, 95% CI 2-sided [-0.17 to 0.17]

16. Secondary Outcome: Influence of Co-morbidities on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction for the injection device. Co-morbidities categories were defined based on current usage of tobacco and alcoholic beverages. Participants were divided into categories, yes and no, for both current tobacco usage and current alcohol usage.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Current tobacco usage: Yes | 8.94 (2.11) | 7.40 (2.60)
  Current tobacco usage: No | 8.95 (1.70) | 7.76 (2.58)
  Current alcohol usage: Yes | 8.96 (1.93) | 8.06 (2.06)
  Current alcohol usage: No | 8.94 (1.84) | 7.33 (2.86)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between categories, current tobacco usage: yes and current tobacco usage: no (reference); Test type: Superiority or Other; p = 0.531, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = -0.15, 95% CI 2-sided [-0.61 to 0.32]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between categories, current alcohol usage: yes and current alcohol usage: no (reference); Test type: Superiority or Other; p = 0.061, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = 0.44, 95% CI 2-sided [-0.02 to 0.90]

17. Secondary Outcome: Influence of Prior Systemic Treatment or Topical Medication for Psoriasis on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the injection device. The categories were defined based on presence of any prior experience of systemic treatment or topical medication for psoriasis. Participants were divided into categories: yes and no.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Yes | 8.95 (1.87) | 7.61 (2.59)
  No | NA (NA) — Data was not analyzed because all the participants had received prior systemic or topical medication. | 9.00 (NA) — Data was not available because there was only 1 participant who did not receive any prior systemic or topical medication.
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between categories, yes and no (reference); Test type: Superiority or Other; p = 0.759, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = -0.73, 95% CI 2-sided [-5.37 to 3.92]

18. Secondary Outcome: Influence of Prior Injection Experience on Participant Satisfaction With Injection Device
Description: Participant satisfaction was scored on a 10-point ordinal scale: 0=totally dissatisfied to 10=totally satisfied. Higher scores indicated greater satisfaction with the injection device. The categories were defined based on presence of any prior experience of injection. Participants were divided into categories: yes and no.
Time Frame: Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Yes | 9.05 (1.66) | 7.70 (2.58)
  No | 8.88 (2.01) | 7.56 (2.61)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Statistical analysis was carried out between categories, yes and no (reference); Test type: Superiority or Other; p = 0.713, Regression, Linear — Statistical testing, 2-sided, was done at 5% significance level; Regression coefficient = 0.09, 95% CI 2-sided [-0.37 to 0.55]

19. Secondary Outcome: Ease of Use of Injection Device Based on Response to Question Concerning Overall Ease in Performing Injection With Device
Description: Ease of use of injection device was assessed by participant's response to question, "How easy was it to perform an injection with this device?" scored on a 5-point Likert scale (0= very easy to 4= very difficult).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 (n=202, 208) | 134 | 92
  Baseline- After the training: 1 (n=202, 208) | 50 | 72
  Baseline- After the training: 2 (n=202, 208) | 15 | 33
  Baseline- After the training: 3 (n=202, 208) | 3 | 7
  Baseline- After the training: 4 (n=202, 208) | 0 | 4
  Week 4: 0 (n=180, 190) | 126 | 94
  Week 4: 1 (n=180, 190) | 42 | 62
  Week 4: 2 (n=180, 190) | 6 | 20
  Week 4: 3 (n=180, 190) | 2 | 12
  Week 4: 4 (n=180, 190) | 4 | 2
  Week 12: 0 (n=194, 195) | 149 | 109
  Week 12: 1 (n=194, 195) | 35 | 54
  Week 12: 2 (n=194, 195) | 4 | 18
  Week 12: 3 (n=194, 195) | 4 | 9
  Week 12: 4 (n=194, 195) | 2 | 5
  Last observation: 0 (n=202, 207) | 153 | 115
  Last observation: 1 (n=202, 207) | 36 | 58
  Last observation: 2 (n=202, 207) | 4 | 19
  Last observation: 3 (n=202, 207) | 5 | 9
  Last observation: 4 (n=202, 207) | 4 | 6
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Baseline- after the training: A GEE model, using a cumulative logit link, a multinomial distribution and an independent correlation structure, with device group, visit and the interaction between device group and visit as fixed factors, was used to analyze individual concepts and questions measuring participant perception; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.39, 95% CI 2-sided [1.63 to 3.49]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Week 4:A GEE model, using a cumulative logit link, a multinomial distribution and an independent correlation structure, with device group, visit and the interaction between device group and visit as fixed factors, was used to analyze individual concepts and questions measuring participant perception; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.61 to 3.67]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Week 12: A GEE model, using a cumulative logit link, a multinomial distribution and an independent correlation structure, with device group, visit and the interaction between device group and visit as fixed factors, was used to analyze individual concepts and questions measuring participant perception; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.74, 95% CI 2-sided [1.78 to 4.21]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Last observation: Logistic regression was used to analyze individual concepts and questions measuring participant perception; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.66 to 3.80]

20. Secondary Outcome: Ease of Use of Injection Device Based on Response to Question Concerning Ease in Learning How to Use Device
Description: Ease of use of injection device was assessed by participant's response to question, "How easy was it to use the device?" scored on a 5-point Likert scale (0= very easy to 4= very difficult).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 (n=201, 208) | 154 | 132
  Baseline- After the training: 1 (n=201, 208) | 39 | 57
  Baseline- After the training: 2 (n=201, 208) | 7 | 13
  Baseline- After the training: 3 (n=201, 208) | 1 | 5
  Baseline- After the training: 4 (n=201, 208) | 0 | 1
  Week 4: 0 (n=179, 189) | 137 | 122
  Week 4: 1 (n=179, 189) | 32 | 54
  Week 4: 2 (n=179, 189) | 4 | 6
  Week 4: 3 (n=179, 189) | 1 | 4
  Week 4: 4 (n=179, 189) | 5 | 3
  Week 12: 0 (n=189, 195) | 154 | 126
  Week 12: 1 (n=189, 195) | 26 | 54
  Week 12: 2 (n=189, 195) | 4 | 9
  Week 12: 3 (n=189, 195) | 2 | 2
  Week 12: 4 (n=189, 195) | 3 | 4
  Last observation: 0 (n=201, 207) | 161 | 134
  Last observation: 1 (n=201, 207) | 26 | 57
  Last observation: 2 (n=201, 207) | 6 | 10
  Last observation: 3 (n=201, 207) | 5 | 2
  Last observation: 4 (n=201, 207) | 3 | 4
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.004, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.22 to 2.89]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Week 4: A GEE model, using a cumulative logit link, a multinomial distribution and an independent correlation structure, with device group, visit and the interaction between device group and visit as fixed factors, was used to analyze individual concepts and questions measuring participant perception; Test type: Superiority or Other; p = 0.017, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.10 to 2.72]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.47 to 3.73]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.32 to 3.21]

21. Secondary Outcome: Ease of Use of Injection Device Based on Response to Question Concerning Ease in Disposing Off Device
Description: Ease of use of injection device was assessed by participant's response to question, "How easy was it to dispose of the device?" scored on a 5-point Likert scale (0= very easy to 4= very difficult).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 (n=198, 205) | 158 | 141
  Baseline- After the training: 1 (n=198, 205) | 25 | 47
  Baseline- After the training: 2 (n=198, 205) | 12 | 9
  Baseline- After the training: 3 (n=198, 205) | 3 | 2
  Baseline- After the training: 4 (n=198, 205) | 0 | 6
  Week 4: 0 (n=173, 189) | 131 | 142
  Week 4: 1 (n=173, 189) | 29 | 34
  Week 4: 2 (n=173, 189) | 5 | 5
  Week 4: 3 (n=173, 189) | 4 | 5
  Week 4: 4 (n=173, 189) | 4 | 3
  Week 12: 0 (n=187, 195) | 150 | 148
  Week 12: 1 (n=187, 195) | 21 | 34
  Week 12: 2 (n=187, 195) | 6 | 9
  Week 12: 3 (n=187, 195) | 4 | 2
  Week 12: 4 (n=187, 195) | 6 | 2
  Last observation: 0 (n=202, 210) | 161 | 161
  Last observation: 1 (n=202, 210) | 23 | 36
  Last observation: 2 (n=202, 210) | 6 | 9
  Last observation: 3 (n=202, 210) | 5 | 2
  Last observation: 4 (n=202, 210) | 7 | 2
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.025, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.07 to 2.64]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.936, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.63 to 1.64]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.420, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.75 to 1.99]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.625, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.71 to 1.79]

22. Secondary Outcome: Ease of Use of Injection Device Based on Response to Question Concerning Ease in Knowing When Injection is Complete
Description: Ease of use of injection device was assessed by participant's response to question, "How easy is it to know when the injection is completed?" scored on a 5-point Likert scale (0= very easy to 4= very difficult).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 (n=201, 207) | 140 | 129
  Baseline- After the training: 1 (n=201, 207) | 44 | 62
  Baseline- After the training: 2 (n=201, 207) | 13 | 10
  Baseline- After the training: 3 (n=201, 207) | 3 | 4
  Baseline- After the training: 4 (n=201, 207) | 1 | 2
  Week 4: 0 (n=175, 189) | 124 | 123
  Week 4: 1 (n=175, 189) | 40 | 50
  Week 4: 2 (n=175, 189) | 5 | 8
  Week 4: 3 (n=175, 189) | 2 | 5
  Week 4: 4 (n=175, 189) | 4 | 3
  Week 12: 0 (n=194, 192) | 147 | 137
  Week 12: 1 (n=194, 192) | 40 | 38
  Week 12: 2 (n=194, 192) | 4 | 9
  Week 12: 3 (n=194, 192) | 0 | 6
  Week 12: 4 (n=194, 192) | 3 | 2
  Last Observation: 0 (n=204, 210) | 155 | 151
  Last Observation: 1 (n=204, 210) | 42 | 42
  Last Observation: 2 (n=204, 210) | 4 | 9
  Last Observation: 3 (n=204, 210) | 0 | 6
  Last Observation: 4 (n=204, 210) | 3 | 2
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.210, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.86 to 1.94]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.227, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.85 to 2.03]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.220, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.84 to 2.08]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.249, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.84 to 2.00]

23. Secondary Outcome: Ease of Use of Injection Device Based on Response to Question Concerning Ease in Holding Device While Injecting
Description: Ease of use of injection device was assessed by participant's response to question, "How easy is it to hold the device whilst injecting?" scored on a 5-point Likert scale (0= very easy to 4= very difficult)
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 (n=199, 206) | 134 | 100
  Baseline- After the training: 1 (n=199, 206) | 48 | 72
  Baseline- After the training: 2 (n=199, 206) | 15 | 24
  Baseline- After the training: 3 (n=199, 206) | 2 | 8
  Baseline- After the training: 4 (n=199, 206) | 0 | 2
  Week 4: 0 (n=179, 190) | 114 | 83
  Week 4: 1 (n=179, 190) | 45 | 59
  Week 4: 2 (n=179, 190) | 14 | 33
  Week 4: 3 (n=179, 190) | 3 | 12
  Week 4: 4 (n=179, 190) | 3 | 3
  Week 12: 0 (n=193, 196) | 133 | 101
  Week 12: 1 (n=193, 196) | 51 | 55
  Week 12: 2 (n=193, 196) | 4 | 27
  Week 12: 3 (n=193, 196) | 1 | 10
  Week 12: 4 (n=193, 196) | 4 | 3
  Last observation: 0 (n=203, 209) | 140 | 105
  Last observation: 1 (n=203, 209) | 52 | 61
  Last observation: 2 (n=203, 209) | 6 | 29
  Last observation: 3 (n=203, 209) | 1 | 11
  Last observation: 4 (n=203, 209) | 4 | 3
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.001, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.48 to 3.21]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.62 to 3.62]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.35, 95% CI 2-sided [1.58 to 3.51]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.64 to 3.59]

24. Secondary Outcome: Ease of Use of Injection Device Based on Response to Question Concerning Hand Discomfort While Injecting
Description: Ease of use of injection device was assessed by participant's response to question, "Did you feel any hand discomfort whilst using the device?" scored on a 5-point Likert scale (0= none to 4= extreme).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 (n=197, 208) | 158 | 131
  Baseline- After the training: 1 (n=197, 208) | 26 | 44
  Baseline- After the training: 2 (n=197, 208) | 6 | 20
  Baseline- After the training: 3 (n=197, 208) | 3 | 10
  Baseline- After the training: 4 (n=197, 208) | 4 | 3
  Week 4: 0 (n=176, 188) | 144 | 114
  Week 4: 1 (n=176, 188) | 18 | 37
  Week 4: 2 (n=176, 188) | 7 | 26
  Week 4: 3 (n=176, 188) | 7 | 8
  Week 4: 4 (n=176, 188) | 0 | 3
  Week 12: 0 (n=193, 195) | 159 | 125
  Week 12: 1 (n=193, 195) | 24 | 45
  Week 12: 2 (n=193, 195) | 7 | 15
  Week 12: 3 (n=193, 195) | 2 | 7
  Week 12: 4 (n=193, 195) | 1 | 3
  Last observation: 0 (n=204, 210) | 168 | 138
  Last observation: 1 (n=204, 210) | 25 | 46
  Last observation: 2 (n=204, 210) | 8 | 15
  Last observation: 3 (n=204, 210) | 2 | 8
  Last observation: 4 (n=204, 210) | 1 | 3
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.001, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.50 to 3.65]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.96, 95% CI 2-sided [1.83 to 4.77]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.58, 95% CI 2-sided [1.62 to 4.12]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.45, 95% CI 2-sided [1.55 to 3.86]

25. Secondary Outcome: Ease of Use of Injection Device Based on Response to Question Concerning Time Taken to Perform Injection (Includes Preparation and Disposal)
Description: Ease of Use of Injection Device was assessed by participant's response to question, "How long does it take to perform the injection, including any preparation and disposal?" where time spent was recorded in minutes and categorized into 5 categories, ranging from 'less than 5 minutes' to 'more than 30 minutes'.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After training: less than 5 (n=200, 206) | 132 | 129
  Baseline- After training: 5 to10 (n=200, 206) | 43 | 56
  Baseline- After training: 11 to 20 (n=200, 206) | 12 | 14
  Baseline- After training: 21 to 30 (n=200, 206) | 9 | 7
  Baseline- After training:more than 30 (n=200, 206) | 4 | 0
  Week 4: less than 5 (n=180, 189) | 117 | 121
  Week 4: 5 to 10 (n=180, 189) | 36 | 41
  Week 4: 11 to 20 (n=180, 189) | 14 | 16
  Week 4: 21 to 30 (n=180, 189) | 8 | 10
  Week 4: more than 30 (n=180, 189) | 5 | 1
  Week 12: less than 5 (n=192, 196) | 124 | 132
  Week 12: 5 to 10 (n=192, 196) | 44 | 40
  Week 12: 11 to 20 (n=192, 196) | 12 | 12
  Week 12: 21 to 30 (n=192, 196) | 6 | 7
  Week 12: more than 30 (n=192, 196) | 6 | 5
  Last observation: less than 5 (n=204, 210) | 131 | 143
  Last observation: 5 to 10 (n=204, 210) | 48 | 43
  Last observation: 11 to 20 (n=204, 210) | 12 | 12
  Last observation: 21 to 30 (n=204, 210) | 7 | 7
  Last observation: more than 30 (n=204, 210) | 6 | 5
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.681, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.73 to 1.62]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.947, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.67 to 1.54]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.604, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.59 to 1.36]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.430, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.57 to 1.27]

26. Secondary Outcome: Convenience of Injection Device Based on Response to Question Concerning Extent of Interference of Injecting Drug With Ability to Enjoy Social or Leisure Activity
Description: Convenience of injection device was assessed by participant's response to question, "How much do you think injecting etanercept will interfere with your ability to enjoy social or leisure activities?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: mITT analysis population included all randomized participants who received at least 1 injection of study medication and had at least 1 efficacy evaluation.
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 116 | 134
  Baseline- After the training: 1 | 34 | 37
  Baseline- After the training: 2 | 30 | 20
  Baseline- After the training: 3 | 11 | 8
  Baseline- After the training: 4 | 12 | 9
  Week 4: 0 | 145 | 138
  Week 4: 1 | 32 | 34
  Week 4: 2 | 6 | 14
  Week 4: 3 | 8 | 8
  Week 4: 4 | 5 | 7
  Week 12: 0 | 133 | 131
  Week 12: 1 | 44 | 33
  Week 12: 2 | 8 | 17
  Week 12: 3 | 4 | 7
  Week 12: 4 | 6 | 9
  Last observation: 0 | 139 | 144
  Last observation: 1 | 46 | 34
  Last observation: 2 | 8 | 17
  Last observation: 3 | 5 | 7
  Last observation: 4 | 8 | 9
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.072, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.48 to 1.03]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.205, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.86 to 2.03]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.434, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.78 to 1.78]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.857, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.69 to 1.55]

27. Secondary Outcome: Convenience of Injection Device Based on Response to Question Concerning Interference of Injecting Drug With Usual Daily Activity
Description: Convenience of injection device was assessed by participant's response to question, "Do you think injecting etanercept will interfere with your usual daily activities?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 134 | 137
  Baseline- After the training: 1 | 45 | 45
  Baseline- After the training: 2 | 14 | 16
  Baseline- After the training: 3 | 6 | 5
  Baseline- After the training: 4 | 3 | 5
  Week 4: 0 | 150 | 145
  Week 4: 1 | 35 | 37
  Week 4: 2 | 4 | 8
  Week 4: 3 | 3 | 7
  Week 4: 4 | 2 | 4
  Week 12: 0 | 147 | 137
  Week 12: 1 | 40 | 39
  Week 12: 2 | 6 | 13
  Week 12: 3 | 0 | 4
  Week 12: 4 | 2 | 5
  Last observation: 0 | 155 | 148
  Last observation: 1 | 42 | 40
  Last observation: 2 | 7 | 13
  Last observation: 3 | 0 | 4
  Last observation: 4 | 2 | 5
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.837, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.70 to 1.56]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.172, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.87 to 2.15]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.096, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.94 to 2.24]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.164, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.88 to 2.08]

28. Secondary Outcome: Convenience of Injection Device Based on Response to Question Concerning Interference of Injecting Drug With Traveling
Description: Convenience of injection device was assessed by participant's response to question, "How much do you think injecting etanercept will interfere with travelling on holiday or business or visiting?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 105 | 98
  Baseline- After the training: 1 | 48 | 55
  Baseline- After the training: 2 | 34 | 32
  Baseline- After the training: 3 | 13 | 20
  Baseline- After the training: 4 | 3 | 3
  Week 4: 0 | 101 | 107
  Week 4: 1 | 46 | 37
  Week 4: 2 | 34 | 33
  Week 4: 3 | 9 | 12
  Week 4: 4 | 3 | 10
  Week 12: 0 | 109 | 101
  Week 12: 1 | 44 | 40
  Week 12: 2 | 33 | 36
  Week 12: 3 | 5 | 12
  Week 12: 4 | 4 | 8
  Last observation: 0 | 115 | 111
  Last observation: 1 | 46 | 43
  Last observation: 2 | 34 | 37
  Last observation: 3 | 7 | 12
  Last observation: 4 | 4 | 8
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.356, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.83 to 1.69]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.737, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.73 to 1.56]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.156, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.90 to 1.91]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.290, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.85 to 1.76]

29. Secondary Outcome: Confidence in Injection Device Based on Response to Question Concerning Overall Confidence in Management of Injections
Description: Confidence in injection device was assessed by participant's response to question, "How confident are you in your management of your injections?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 6 | 11
  Baseline- After the training: 1 | 13 | 20
  Baseline- After the training: 2 | 30 | 31
  Baseline- After the training: 3 | 76 | 78
  Baseline- After the training: 4 | 81 | 67
  Week 4: 0 | 4 | 3
  Week 4: 1 | 9 | 8
  Week 4: 2 | 6 | 10
  Week 4: 3 | 56 | 75
  Week 4: 4 | 121 | 105
  Week 12: 0 | 9 | 1
  Week 12: 1 | 5 | 7
  Week 12: 2 | 7 | 12
  Week 12: 3 | 47 | 60
  Week 12: 4 | 131 | 117
  Last observation: 0 | 9 | 2
  Last observation: 1 | 5 | 7
  Last observation: 2 | 7 | 13
  Last observation: 3 | 49 | 67
  Last observation: 4 | 136 | 122
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.065, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.50 to 1.02]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.100, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.50 to 1.06]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.298, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.54 to 1.21]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.148, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.51 to 1.11]

30. Secondary Outcome: Confidence in Injection Device Based on Response to Question Concerning Confidence That Participant Injects Right Amount of Drug Every Time
Description: Confidence in injection device was assessed by participant's response to question, "How confident are you that you inject the right amount of medicine every time?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 5 | 2
  Baseline- After the training: 1 | 4 | 7
  Baseline- After the training: 2 | 19 | 15
  Baseline- After the training: 3 | 67 | 54
  Baseline- After the training: 4 | 111 | 129
  Week 4: 0 | 5 | 3
  Week 4: 1 | 3 | 6
  Week 4: 2 | 8 | 3
  Week 4: 3 | 53 | 50
  Week 4: 4 | 126 | 139
  Week 12: 0 | 7 | 2
  Week 12: 1 | 4 | 6
  Week 12: 2 | 7 | 7
  Week 12: 3 | 48 | 43
  Week 12: 4 | 132 | 139
  Last observation: 0 | 7 | 3
  Last observation: 1 | 4 | 6
  Last observation: 2 | 8 | 7
  Last observation: 3 | 52 | 47
  Last observation: 4 | 135 | 148
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.098, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.94 to 2.03]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.311, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.82 to 1.87]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.376, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.79 to 1.85]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.299, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.83 to 1.86]

31. Secondary Outcome: Confidence in Injection Device Based on Response to Question Concerning Confidence That Participant Can Inject Properly With Device
Description: Confidence in injection device was assessed by participant's response to question, "How confident are you that you can inject yourself properly with the device?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 4 | 2
  Baseline- After the training: 1 | 3 | 7
  Baseline- After the training: 2 | 12 | 27
  Baseline- After the training: 3 | 70 | 53
  Baseline- After the training: 4 | 117 | 116
  Week 4: 0 | 6 | 3
  Week 4: 1 | 0 | 5
  Week 4: 2 | 7 | 10
  Week 4: 3 | 47 | 65
  Week 4: 4 | 135 | 118
  Week 12: 0 | 9 | 1
  Week 12: 1 | 1 | 6
  Week 12: 2 | 4 | 12
  Week 12: 3 | 43 | 54
  Week 12: 4 | 142 | 123
  Last observation: 0 | 9 | 2
  Last observation: 1 | 1 | 6
  Last observation: 2 | 4 | 13
  Last observation: 3 | 47 | 60
  Last observation: 4 | 145 | 130
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.494, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.60 to 1.28]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.036, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.44 to 0.97]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.079, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.45 to 1.04]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.063, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.46 to 1.02]

32. Secondary Outcome: Confidence in Injection Device Based on Response to Question Concerning Confidence Regarding Control Over Injection Process
Description: Confidence in injection device was assessed by participant's response to question, "Are you confident that you have good control over the injection process?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 4 | 2
  Baseline- After the training: 1 | 2 | 10
  Baseline- After the training: 2 | 11 | 21
  Baseline- After the training: 3 | 72 | 56
  Baseline- After the training: 4 | 113 | 117
  Week 4: 0 | 3 | 3
  Week 4: 1 | 3 | 4
  Week 4: 2 | 8 | 9
  Week 4: 3 | 49 | 62
  Week 4: 4 | 131 | 122
  Week 12: 0 | 6 | 2
  Week 12: 1 | 3 | 5
  Week 12: 2 | 6 | 10
  Week 12: 3 | 43 | 52
  Week 12: 4 | 141 | 127
  Last observation: 0 | 6 | 2
  Last observation: 1 | 3 | 5
  Last observation: 2 | 8 | 10
  Last observation: 3 | 45 | 59
  Last observation: 4 | 144 | 135
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.628, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.62 to 1.33]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.203, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.51 to 1.15]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.222, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.51 to 1.17]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.263, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.53 to 1.19]

33. Secondary Outcome: Confidence in Injection Device Based on Response to Question Concerning Confidence Regarding Successful Injection
Description: Confidence in injection device was assessed by participant's response to question, "How confident are you that you injected yourself successfully?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 3 | 1
  Baseline- After the training: 1 | 2 | 8
  Baseline- After the training: 2 | 16 | 22
  Baseline- After the training: 3 | 69 | 54
  Baseline- After the training: 4 | 115 | 122
  Week 4: 0 | 3 | 2
  Week 4: 1 | 3 | 3
  Week 4: 2 | 5 | 12
  Week 4: 3 | 60 | 52
  Week 4: 4 | 124 | 132
  Week 12: 0 | 5 | 2
  Week 12: 1 | 3 | 4
  Week 12: 2 | 1 | 10
  Week 12: 3 | 55 | 49
  Week 12: 4 | 135 | 132
  Last observation: 0 | 5 | 2
  Last observation: 1 | 3 | 4
  Last observation: 2 | 2 | 12
  Last observation: 3 | 58 | 53
  Last observation: 4 | 138 | 140
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.914, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.70 to 1.50]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.827, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.70 to 1.57]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.712, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.61 to 1.40]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.733, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.62 to 1.39]

34. Secondary Outcome: Assessment of Fear of Device Based on Response to Question Concerning Nervousness About Injections
Description: Fear of Device was assessed by participant's response to question, "How nervous do you feel about your injections?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 92 | 80
  Baseline- After the training: 1 | 59 | 54
  Baseline- After the training: 2 | 29 | 39
  Baseline- After the training: 3 | 16 | 24
  Baseline- After the training: 4 | 10 | 10
  Week 4: 0 | 110 | 103
  Week 4: 1 | 54 | 51
  Week 4: 2 | 22 | 27
  Week 4: 3 | 7 | 15
  Week 4: 4 | 3 | 5
  Week 12: 0 | 125 | 111
  Week 12: 1 | 53 | 46
  Week 12: 2 | 17 | 19
  Week 12: 3 | 4 | 15
  Week 12: 4 | 0 | 7
  Last observation: 0 | 131 | 119
  Last observation: 1 | 53 | 48
  Last observation: 2 | 18 | 22
  Last observation: 3 | 4 | 15
  Last observation: 4 | 0 | 7
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.090, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.95 to 1.95]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.154, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.90 to 1.91]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.037, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.02 to 2.22]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.028, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.05 to 2.24]

35. Secondary Outcome: Assessment of Fear of Device Based on Response to Question Concerning Nervousness About Inserting Needle Into Skin
Description: Fear of Device was assessed by participant's response to question, "How nervous do you feel about inserting the needle into your skin?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 102 | 82
  Baseline- After the training: 1 | 44 | 49
  Baseline- After the training: 2 | 32 | 38
  Baseline- After the training: 3 | 17 | 22
  Baseline- After the training: 4 | 10 | 16
  Week 4: 0 | 110 | 93
  Week 4: 1 | 61 | 54
  Week 4: 2 | 13 | 29
  Week 4: 3 | 10 | 18
  Week 4: 4 | 1 | 7
  Week 12: 0 | 115 | 105
  Week 12: 1 | 59 | 47
  Week 12: 2 | 19 | 19
  Week 12: 3 | 6 | 19
  Week 12: 4 | 0 | 7
  Last observation: 0 | 121 | 112
  Last observation: 1 | 59 | 52
  Last observation: 2 | 20 | 20
  Last observation: 3 | 6 | 20
  Last observation: 4 | 0 | 7
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.022, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.06 to 2.21]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.005, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.17 to 2.41]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.076, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.97 to 2.03]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.049, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.00 to 2.11]

36. Secondary Outcome: Assessment of Fear of Device Based on Response to Question Concerning Dislike Towards Injecting With Device
Description: Fear of Device was assessed by participant's response to question, "Do you dislike injecting yourself with this device?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 129 | 103
  Baseline- After the training: 1 | 43 | 40
  Baseline- After the training: 2 | 22 | 29
  Baseline- After the training: 3 | 10 | 22
  Baseline- After the training: 4 | 2 | 12
  Week 4: 0 | 135 | 96
  Week 4: 1 | 42 | 52
  Week 4: 2 | 15 | 33
  Week 4: 3 | 0 | 11
  Week 4: 4 | 2 | 9
  Week 12: 0 | 143 | 112
  Week 12: 1 | 39 | 39
  Week 12: 2 | 13 | 28
  Week 12: 3 | 1 | 11
  Week 12: 4 | 3 | 7
  Last observation: 0 | 150 | 119
  Last observation: 1 | 39 | 43
  Last observation: 2 | 13 | 30
  Last observation: 3 | 1 | 12
  Last observation: 4 | 3 | 7
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.001, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.32 to 2.83]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.63, 95% CI 2-sided [1.78 to 3.87]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.42 to 3.19]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 2.27, 95% CI 2-sided [1.52 to 3.39]

37. Secondary Outcome: Assessment of Fear of Device Based on Response to Question Concerning Emotional Distress or Anxiety About Injection
Description: Fear of Device was assessed by participant's response to question, "Are you emotionally distressed or anxious about your injections?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 124 | 105
  Baseline- After the training: 1 | 45 | 57
  Baseline- After the training: 2 | 28 | 26
  Baseline- After the training: 3 | 7 | 11
  Baseline- After the training: 4 | 2 | 7
  Week 4: 0 | 124 | 119
  Week 4: 1 | 57 | 50
  Week 4: 2 | 11 | 21
  Week 4: 3 | 2 | 9
  Week 4: 4 | 1 | 2
  Week 12: 0 | 143 | 125
  Week 12: 1 | 41 | 42
  Week 12: 2 | 12 | 24
  Week 12: 3 | 1 | 5
  Week 12: 4 | 1 | 2
  Last observation: 0 | 149 | 134
  Last observation: 1 | 42 | 45
  Last observation: 2 | 13 | 25
  Last observation: 3 | 1 | 5
  Last observation: 4 | 1 | 2
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.057, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.99 to 2.11]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.151, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.90 to 1.96]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.024, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.06 to 2.44]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.025, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.06 to 2.39]

38. Secondary Outcome: Device Characteristics Based on Response to Question Concerning Look of Device
Description: Device characteristics were assessed by participant's response to question, "How much do you like the look of the device?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 4 | 18
  Baseline- After the training: 1 | 10 | 21
  Baseline- After the training: 2 | 62 | 90
  Baseline- After the training: 3 | 81 | 56
  Baseline- After the training: 4 | 49 | 20
  Week 4: 0 | 3 | 14
  Week 4: 1 | 2 | 22
  Week 4: 2 | 51 | 92
  Week 4: 3 | 79 | 46
  Week 4: 4 | 58 | 27
  Week 12: 0 | 1 | 13
  Week 12: 1 | 11 | 20
  Week 12: 2 | 43 | 77
  Week 12: 3 | 78 | 59
  Week 12: 4 | 66 | 29
  Last observation: 0 | 1 | 14
  Last observation: 1 | 11 | 21
  Last observation: 2 | 46 | 82
  Last observation: 3 | 79 | 62
  Last observation: 4 | 69 | 32
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.001, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.24 to 0.49]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.18 to 0.37]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.31, 95% CI 2-sided [0.21 to 0.45]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.23 to 0.47]

39. Secondary Outcome: Device Characteristics Based on Response to Question Concerning Feel of Device
Description: Device characteristics were assessed by participant's response to question, "How much do you like the feel of the device?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 1 | 9
  Baseline- After the training: 1 | 9 | 24
  Baseline- After the training: 2 | 69 | 92
  Baseline- After the training: 3 | 78 | 60
  Baseline- After the training: 4 | 49 | 19
  Week 4: 0 | 2 | 15
  Week 4: 1 | 7 | 21
  Week 4: 2 | 58 | 90
  Week 4: 3 | 71 | 45
  Week 4: 4 | 55 | 30
  Week 12: 0 | 4 | 7
  Week 12: 1 | 9 | 19
  Week 12: 2 | 46 | 87
  Week 12: 3 | 76 | 54
  Week 12: 4 | 64 | 31
  Last observation: 0 | 4 | 7
  Last observation: 1 | 9 | 20
  Last observation: 2 | 49 | 94
  Last observation: 3 | 77 | 58
  Last observation: 4 | 67 | 32
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.001, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.27 to 0.54]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.31, 95% CI 2-sided [0.21 to 0.46]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.24 to 0.50]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.24 to 0.50]

40. Secondary Outcome: Device Characteristics Based on Response to Question Regarding Comfort to Use Device Based on Looks
Description: Device characteristics were assessed by participant's response to question, "How much does the device look like something you would feel comfortable to use?" scored on a 5-point Likert scale (0= not at all to 4= very much).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the training: 0 | 7 | 32
  Baseline- After the training: 1 | 11 | 26
  Baseline- After the training: 2 | 68 | 76
  Baseline- After the training: 3 | 67 | 55
  Baseline- After the training: 4 | 53 | 16
  Week 4: 0 | 6 | 28
  Week 4: 1 | 8 | 22
  Week 4: 2 | 51 | 74
  Week 4: 3 | 69 | 45
  Week 4: 4 | 59 | 32
  Week 12: 0 | 7 | 27
  Week 12: 1 | 15 | 21
  Week 12: 2 | 47 | 62
  Week 12: 3 | 65 | 54
  Week 12: 4 | 65 | 34
  Last observation: 0 | 7 | 27
  Last observation: 1 | 16 | 22
  Last observation: 2 | 47 | 68
  Last observation: 3 | 67 | 58
  Last observation: 4 | 69 | 36
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p < 0.001, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.24 to 0.46]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.22 to 0.46]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.26 to 0.56]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.28 to 0.58]

41. Secondary Outcome: Side Effects Related to Administration Based on Response to Question Concerning Experience of Pain During or Immediately After Injection
Description: Side effects related to administration were assessed by participant's response to question, "Do you experience pain during or immediately after the injection?" scored on a 5-point Likert scale (0= none to 4= severe).
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Baseline- After the first injection: 0 | 98 | 109
  Baseline- After the first injection: 1 | 65 | 54
  Baseline- After the first injection: 2 | 24 | 31
  Baseline- After the first injection: 3 | 9 | 8
  Baseline- After the first injection: 4 | 3 | 0
  Week 4: 0 | 77 | 88
  Week 4: 1 | 60 | 60
  Week 4: 2 | 33 | 31
  Week 4: 3 | 22 | 21
  Week 4: 4 | 3 | 1
  Week 12: 0 | 76 | 84
  Week 12: 1 | 68 | 70
  Week 12: 2 | 30 | 28
  Week 12: 3 | 21 | 15
  Week 12: 4 | 4 | 1
  Last observation: 0 | 79 | 90
  Last observation: 1 | 70 | 72
  Last observation: 2 | 31 | 32
  Last observation: 3 | 22 | 16
  Last observation: 4 | 4 | 1
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Baseline- after the first injection: A GEE model, using a cumulative logit link, a multinomial distribution and an independent correlation structure, with device group, visit and the interaction between device group and visit as fixed factors, was used to analyze individual concepts and questions measuring participant perception; Test type: Superiority or Other; p = 0.470, Generalized estimating equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.60 to 1.26]
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 20, analysis 2]; Test type: Superiority or Other; p = 0.325, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.57 to 1.20]
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.197, Generalized Estimating Equations — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.55 to 1.13]
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 19, analysis 4]; Test type: Superiority or Other; p = 0.212, Regression, Logistic — Statistical testing, 2-sided, was done at 5% significance level; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.56 to 1.14]

42. Secondary Outcome: Short Form State-Trait Anxiety Inventory (SF STAI) Global Score
Description: SF-STAI is a 6 item short form. Global score = sum of coded answers/number of answered questions multiplied by 6, with answers coded on a 4 point Likert scale, where 1 = least anxious and 4 = most anxious. The global score ranges from 6 to 24, where higher score shows greater anxiety.
Time Frame: Baseline, Week 4 and Week 12
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Baseline- After the training | 11.0 (3.5) | 11.2 (3.6)
  Week 4 | 9.9 (3.3) | 10.0 (3.5)
  Week 12 | 10.1 (3.2) | 10.1 (3.3)
  Last observation | 10.1 (3.3) | 10.1 (3.3)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Baseline- after the training: Mixed linear model with participant as random effect, treatment group, visit and the interaction between treatment group and visit as fixed factors and with an auto-regressive correlation structure was used to calculate 95% CI; Test type: Superiority or Other; p = 0.515, ANOVA — Statistical testing, 2-sided, was done at 5% significance level; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.91 to 0.46], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Week 4: Mixed linear model with participant as random effect, treatment group, visit and the interaction between treatment group and visit as fixed factors and with an unstructured correlation was used for the analysis; Test type: Superiority or Other; p = 0.842, ANOVA — Statistical testing, 2-sided, was done at 5% significance level; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.74 to 0.60], Standard Error of Mean 0.34
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Week 12: Mixed linear model with participant as random effect, treatment group, visit and the interaction between treatment group and visit as fixed factors and with an unstructured correlation was used for the analysis; Test type: Superiority or Other; p = 0.928, ANOVA — Statistical testing, 2-sided, was done at 5% significance level; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.67 to 0.61], Standard Error of Mean 0.33
Statistical Analysis 4: Comparison: Etanercept 50 mg Auto-injector vs Etanercept 50 mg Prefilled Syringe; Last observation: ANOVA method was used for the analysis; Test type: Superiority or Other; p = 0.974, ANOVA — Statistical testing, 2-sided, was done at 5% significance level; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.62 to 0.64], Standard Error of Mean 0.32

43. Secondary Outcome: Influence of Age on Participant Perception
Description: Participant perception was assessed with the 26 questions of the device attribute and participant questionnaire. Based on the scores assigned to the 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using a multiple correspondence analysis and an ascending hierarchical classification. The age was determined for each cluster of participants.
Time Frame: Baseline
Population: mITT analysis population included all randomized participants who received at least 1 injection of study medication and had at least 1 efficacy evaluation. 'n' is signifying those participants who were evaluated for this measure at the satisfaction level for each group respectively.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
years
  Very satisfied (n=119, 92) | 47.9 (12.6) | 49.1 (12.7)
  Satisfied (n= 56, 65) | 42.8 (12.9) | 43.9 (13.3)
  Less satisfied (n= 20, 41) | 42.7 (15.4) | 42.5 (14.4)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated using ANOVA; Test type: Superiority or Other; p = 0.030, ANOVA
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; p-value for statistical difference between all categories in the etanercept 50 mg prefilled syringe group was calculated using ANOVA; Test type: Superiority or Other; p = 0.010, ANOVA

44. Secondary Outcome: Influence of Gender on Participant Perception
Description: Participant perception was assessed with the 26 questions of the device attribute and participant questionnaire. Based on the scores assigned to the 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using a multiple correspondence analysis and an ascending hierarchical classification. Number of female and male participants was determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Very satisfied: Male (n=119, 92) | 77 | 67
  Very satisfied: Female (n=119, 92) | 42 | 25
  Satisfied: Male (n= 56, 65) | 37 | 45
  Satisfied: Female (n= 56, 65) | 19 | 20
  Less satisfied: Male (n= 20, 41) | 13 | 26
  Less satisfied: Female (n= 20, 41) | 7 | 15
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.984, Chi-squared
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; p-value for statistical difference between all categories in the etanercept 50 mg prefilled syringe group was calculated; Test type: Superiority or Other; p = 0.549, Chi-squared

45. Secondary Outcome: Influence of Socio-educational Status on Participant Perception
Description: Participant perception was assessed with the 26 questions of the device attribute and participant questionnaire. Based on the scores assigned to the 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using a multiple correspondence analysis and an ascending hierarchical classification. Number of participants corresponding to each socio-educational level (reading or writing, high school or baccalaureate level, university level) was determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Very satisfied: Reading/Writing level (n=119, 92) | 41 | 32
  Very satisfied: High school level (n=119, 92) | 56 | 43
  Very satisfied: University level (n=119, 92) | 22 | 17
  Satisfied: Reading/Writing level (n= 56, 65) | 12 | 19
  Satisfied: High school level (n= 56, 65) | 34 | 32
  Satisfied: University level (n= 56, 65) | 10 | 14
  Less satisfied: Reading/Writing level (n= 20, 41) | 10 | 16
  Less satisfied: High school level (n= 20, 41) | 7 | 16
  Less satisfied: University level (n= 20, 41) | 3 | 9
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.158, Fisher Exact
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.808, Chi-squared

46. Secondary Outcome: Influence of Psychological Status Assessed by Hospital Anxiety Depression (HAD) Score on Participant Perception
Description: Participant perception: assessed with the 26 questions of the device attribute and participant questionnaire. Based on the scores assigned to 26 questions, participants were divided into 3 clusters (very satisfied, satisfied, less satisfied) using multiple correspondence analysis and an ascending hierarchical classification. Psychological status: assessed using participant rated questionnaire with 2 subscales for anxiety (HAD-A) and depression (HAD-D). Total score: 0 to 21 for each subscale; higher score = greater severity of symptoms. HAD score was determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Very satisfied: HAD-A (n=119, 92) | 7.0 (3.8) [0.0 to 17.0] | 6.0 (4.6) [0.0 to 19.0]
  Very satisfied: HAD-D (n=119, 92) | 5.0 (3.7) [0.0 to 18.0] | 4.0 (3.9) [0.0 to 16.0]
  Satisfied: HAD-A (n= 56, 65) | 7.0 (4.3) [2.0 to 20.0] | 7.0 (4.1) [0.0 to 16.0]
  Satisfied: HAD-D (n= 56, 65) | 5.5 (4.0) [0.0 to 17.0] | 5.0 (3.3) [0.0 to 14.0]
  Less satisfied: HAD-A (n= 20, 41) | 9.2 (3.5) [3.0 to 16.0] | 10.0 (4.2) [2.0 to 17.0]
  Less satisfied: HAD-D (n= 20, 41) | 6.5 (4.2) [0.0 to 14.0] | 8.0 (4.0) [0.0 to 15.0]
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between categories, very satisfied: HAD-A, satisfied: HAD-A and less satisfied: HAD-A, in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.029, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; p-value for statistical difference between categories, very satisfied: HAD-A, satisfied: HAD-A and less satisfied: HAD-A, in the etanercept 50 mg prefilled syringe group was calculated; Test type: Superiority or Other; p = 0.005, Kruskal-Wallis
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between categories, very satisfied: HAD-D, satisfied: HAD-D and less satisfied: HAD-D, in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.411, Kruskal-Wallis
Statistical Analysis 4: Comparison: Etanercept 50 mg Prefilled Syringe; p-value for statistical difference between categories, very satisfied: HAD-D, satisfied: HAD-D and less satisfied: HAD-D, in the etanercept 50 mg prefilled syringe group was calculated; Test type: Superiority or Other; p = 0.005, Kruskal-Wallis

47. Secondary Outcome: Influence of Willingness to Self Manage Assessed by Patient Activation Measure (PAM) on Participant Perception
Description: Participant perception: assessed with 26 questions of device attribute and participant questionnaire. Based on scores assigned to 26 questions, participants were divided into 3 clusters (very satisfied, satisfied, less satisfied) using multiple correspondence analysis and ascending hierarchical classification. The 13-item short form of PAM survey assessed participants' knowledge, skill, and confidence for self-management; score range 0 to 100. Higher scores indicated more confidence in managing participants' condition and lifestyle. PAM score was determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Very satisfied (n=116, 91) | 58.0 (13.8) | 60.5 (14.0)
  Satisfied (n= 56, 63) | 53.0 (11.7) | 57.5 (11.8)
  Less satisfied (n= 20, 40) | 60.0 (13.9) | 52.4 (12.6)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.039, ANOVA
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.006, ANOVA

48. Secondary Outcome: Influence of Prior Injection Experience on Participant Perception
Description: Participant perception was assessed with the 26 questions of the device attribute and participant questionnaire. Based on the scores assigned to the 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using a multiple correspondence analysis and an ascending hierarchical classification. Numbers of participants with and without prior injection experience were determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Very satisfied: with experience (n=119, 92) | 47 | 43
  Very satisfied: without experience (n=119, 92) | 72 | 49
  Satisfied: with experience (n= 56, 65) | 20 | 28
  Satisfied: without experience (n= 56, 65) | 36 | 37
  Less satisfied: with experience (n= 20, 41) | 9 | 16
  Less satisfied: without experience (n= 20, 41) | 11 | 25
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.752, Chi-squared
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.700, Chi-squared

49. Secondary Outcome: Influence of Prior Self-injection Experience on Participant Perception
Description: Participant perception was assessed with the 26 questions of the device attribute and participant questionnaire. Based on the scores assigned to the 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using a multiple correspondence analysis and an ascending hierarchical classification. Numbers of participants with and without prior self-injection experience were determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Very satisfied: with experience (n=119, 92) | 23 | 33
  Very satisfied: without experience (n=119, 92) | 96 | 59
  Satisfied: with experience (n= 56, 65) | 13 | 16
  Satisfied: without experience (n= 56, 65) | 43 | 49
  Less satisfied: with experience (n= 20, 41) | 5 | 9
  Less satisfied: without experience (n= 20, 41) | 15 | 32
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.697, Fisher Exact
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.159, Chi-squared

50. Secondary Outcome: Influence of Duration of Psoriasis on Participant Perception
Description: Participant perception was assessed with the 26 questions of the device attribute and participant questionnaire. Based on the scores assigned to the 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using a multiple correspondence analysis and an ascending hierarchical classification. The duration of psoriasis was determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
years
  Very satisfied (n=119, 92) | 23.3 (13.3) [1.0 to 61.0] | 22.9 (12.1) [1.0 to 63.0]
  Satisfied (n= 56, 65) | 17.8 (10.0) [3.0 to 41.0] | 20.6 (10.8) [2.0 to 53.0]
  Less satisfied (n= 20, 41) | 16.1 (7.4) [4.0 to 30.0] | 17.1 (9.8) [3.0 to 46.0]
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.004, ANOVA
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.024, ANOVA

51. Secondary Outcome: Influence of Physician Global Assessment (PGA) of Psoriasis on Participant Perception
Description: Participant perception was assessed with the 26 questions of the device attribute and participant questionnaire. Based on the scores assigned to the 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using a multiple correspondence analysis and an ascending hierarchical classification. PGA of psoriasis scale ranges from 0 (no psoriasis) to 5 (severe disease). 'Clear' and 'Almost clear' includes all participants who were scored as a 0 or 1. The PGA score was determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Very satisfied (n=119, 92) | 3.0 (0.8) [1.0 to 5.0] | 3.0 (0.6) [2.0 to 5.0]
  Satisfied (n= 56, 65) | 3.0 (0.7) [2.0 to 5.0] | 3.0 (0.8) [1.0 to 5.0]
  Less satisfied (n= 20, 40) | 3.0 (0.7) [2.0 to 5.0] | 3.0 (0.8) [1.0 to 5.0]
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.652, Kruskal-Wallis
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.024, Kruskal-Wallis

52. Secondary Outcome: Influence of Psoriasis Area Severity Index (PASI) on Participant Perception
Description: Participant perception:assessed with 26 questions of device attribute and participant questionnaire. Based on scores assigned to 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using multiple correspondence analysis and ascending hierarchical classification. PASI: combined assessment of lesion severity and area affected into single score; range: 0=no disease to 72=maximal disease. While assessing, body was divided into 4 sections: head, upper extremities, trunk, lower extremities. PASI score was determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Very satisfied (n=118, 92) | 17.2 (7.5) | 17.9 (8.5)
  Satisfied (n= 56, 65) | 18.6 (9.8) | 17.5 (7.9)
  Less satisfied (n= 20, 39) | 17.1 (8.0) | 15.9 (10.2)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.560, ANOVA
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.474, ANOVA

53. Secondary Outcome: Influence of Participant's Assessment of General Health on Participant Perception
Description: Participant perception: assessed with 26 questions of device attribute and participant questionnaire. Based on scores assigned to 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using multiple correspondence analysis and ascending hierarchical classification. Participant's assessment of general health was measured on 100mm line visual analog scale (VAS). 0mm = extremely bad to 100mm = very well. The participant's assessment of general health score was determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
mm
  Very satisfied (n=117, 90) | 64.9 (23.7) | 63.8 (27.9)
  Satisfied (n= 55, 65) | 59.3 (25.3) | 70.7 (21.5)
  Less satisfied (n= 20, 40) | 48.8 (31.2) | 60.5 (22.7)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.023, ANOVA
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.089, ANOVA

54. Secondary Outcome: Influence of Participant's Global Assessment of Psoriasis on Participant Perception
Description: Participant perception: assessed with 26 questions of device attribute and participant questionnaire. Based on scores assigned to 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using multiple correspondence analysis and ascending hierarchical classification. Participant's global assessment of psoriasis was measured using a 100 mm VAS, with 0 = no activity and 100 = extremely active psoriasis. The participant's assessment of psoriasis score was determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
mm
  Very satisfied (n=116, 90) | 73.5 (17.7) | 73.4 (18.0)
  Satisfied (n= 55, 65) | 69.9 (19.1) | 73.3 (19.8)
  Less satisfied (n= 20, 39) | 72.6 (21.2) | 70.8 (26.7)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.494, ANOVA
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.782, ANOVA

55. Secondary Outcome: Influence of Dermatology Life Quality Index (DLQI) on Participant Perception
Description: Participant perception: assessed with 26 questions of device attribute and participant questionnaire. Based on scores assigned to 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using multiple correspondence analysis and ascending hierarchical classification. DLQI is the dermatology-specific quality of life measure used for psoriatic population. The 10-item questionnaire has a score range of 0 to 30 with higher scores indicating poor quality of life. The DLQI score was determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
units on a scale
  Very satisfied (n=116, 90) | 13.4 (6.8) | 13.1 (7.1)
  Satisfied (n= 54, 63) | 12.4 (6.4) | 12.8 (6.0)
  Less satisfied (n= 18, 41) | 14.6 (6.9) | 13.1 (6.7)
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between all categories in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.444, ANOVA
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.947, ANOVA

56. Secondary Outcome: Influence of Co-morbidities on Participant Perception
Description: Participant perception: assessed with 26 questions of device attribute and participant questionnaire. Based on scores assigned to 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using multiple correspondence analysis and ascending hierarchical classification. Co-morbidities included current usage of tobacco and alcoholic beverages. Numbers of participants with and without co-morbidities were determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Very satisfied: Tobacco usage- Yes (n=119, 92) | 49 | 31
  Very satisfied: Tobacco usage- No (n=119, 92) | 70 | 61
  Very satisfied: Alcohol usage- Yes (n=119, 92) | 59 | 38
  Very satisfied: Alcohol usage- No (n=119, 92) | 60 | 54
  Satisfied: Tobacco usage- Yes (n= 56, 65) | 20 | 25
  Satisfied: Tobacco usage- No (n= 56, 65) | 36 | 40
  Satisfied: Alcohol usage- Yes (n= 56, 65) | 20 | 29
  Satisfied: Alcohol usage- No (n= 56, 65) | 36 | 36
  Less satisfied: Tobacco usage- Yes (n= 20, 41) | 8 | 19
  Less satisfied: Tobacco usage- No (n= 20, 41) | 12 | 22
  Less satisfied: Alcohol usage- Yes (n= 20, 41) | 6 | 11
  Less satisfied: Alcohol usage- No (n= 20, 41) | 14 | 30
Statistical Analysis 1: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between categories, very satisfied: tobacco usage- yes, very satisfied: tobacco usage- no, satisfied: tobacco usage- yes, satisfied: tobacco usage- no, less satisfied: tobacco usage- yes and less satisfied: tobacco usage- no, in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.787, Chi-squared
Statistical Analysis 2: Comparison: Etanercept 50 mg Prefilled Syringe; p-value for statistical difference between categories, very satisfied: tobacco usage- yes, very satisfied: tobacco usage- no, satisfied: tobacco usage- yes, satisfied: tobacco usage- no, less satisfied: tobacco usage- yes and less satisfied: tobacco usage- no, in the etanercept 50 mg prefilled syringe group was calculated; Test type: Superiority or Other; p = 0.379, Chi-squared
Statistical Analysis 3: Comparison: Etanercept 50 mg Auto-injector; p-value for statistical difference between categories, very satisfied: alcohol usage- yes, very satisfied: alcohol usage- no, satisfied: alcohol usage- yes, satisfied: alcohol usage- no, less satisfied: alcohol usage- yes and less satisfied: alcohol usage- no, in the etanercept 50 mg auto-injector group was calculated; Test type: Superiority or Other; p = 0.098, Chi-squared
Statistical Analysis 4: Comparison: Etanercept 50 mg Prefilled Syringe; p-value for statistical difference between categories, very satisfied: alcohol usage- yes, very satisfied: alcohol usage- no, satisfied: alcohol usage- yes, satisfied: alcohol usage- no, less satisfied: alcohol usage- yes and less satisfied: alcohol usage- no, in the etanercept 50 mg prefilled syringe group was calculated; Test type: Superiority or Other; p = 0.166, Chi-squared

57. Secondary Outcome: Influence of Prior Systemic Treatment or Topical Medication for Psoriasis on Participant Perception
Description: Participant perception was assessed with the 26 questions of the device attribute and participant questionnaire. Based on the scores assigned to the 26 questions, participants were divided into 3 clusters (very satisfied, satisfied and less satisfied) using a multiple correspondence analysis and an ascending hierarchical classification. Numbers of participants with and without prior experience of systemic or topical treatment for psoriasis were determined for each cluster of participants.
Time Frame: Baseline
Population: as for outcome 43
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Number analyzed (Participants) | 206 | 211
participants
  Very satisfied: Prior medication- Yes (n=119, 92) | 119 | 92
  Very satisfied: Prior medication- No (n=119, 92) | 0 | 0
  Satisfied: Prior medication- Yes (n= 56, 65) | 56 | 64
  Satisfied: Prior medication- No (n= 56, 65) | 0 | 1
  Less satisfied: Prior medication- Yes (n= 20, 41) | 20 | 41
  Less satisfied: Prior medication- No (n= 20, 41) | 0 | 0
Statistical Analysis 1: Comparison: Etanercept 50 mg Prefilled Syringe; [analysis description as in outcome 44, analysis 2]; Test type: Superiority or Other; p = 0.535, Fisher Exact

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept 50 mg Auto-injector | Etanercept 50 mg Prefilled Syringe
Serious Adverse Events (participants affected / at risk) | 6/207 | 5/211
Other Adverse Events (participants affected / at risk) | 94/207 | 96/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept 50 mg Auto-injector (N=207) | Etanercept 50 mg Prefilled Syringe (N=211)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Retinal operation (Surgical and medical procedures) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary calculus removal (Surgical and medical procedures) | 0 | 1
Joint abscess (Infections and infestations) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Prostatic operation (Surgical and medical procedures) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept 50 mg Auto-injector (N=207) | Etanercept 50 mg Prefilled Syringe (N=211)
Injection site erythema (General disorders) | 10 | 17
Injection site haematoma (General disorders) | 10 | 3
Injection site irritation (General disorders) | 6 | 9
Injection site pain (General disorders) | 10 | 10
Injection site pruritis (General disorders) | 3 | 5
Injection site reaction (General disorders) | 18 | 17
Influenza (Infections and infestations) | 5 | 9
Nasopharyngitis (Infections and infestations) | 24 | 27
Upper respiratory tract infection (Infections and infestations) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Headache (Nervous system disorders) | 13 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Erythema (Skin and subcutaneous tissue disorders) | 4 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 13 | 6
Psoriasis (Skin and subcutaneous tissue disorders) | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.